CLINICAL TRIAL: NCT03226535
Title: Ultrasound-CT Fusion System for Interventional Radiology Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clear Guide Medical (Industry)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CGM 17-001
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: CT Guided Biopsy; CT Guided Drain Placement Within the Abdomen or Pelvis; CT Guided Injection of Muscle or Nerve Within the Pelvis
Keywords: Computer Assisted Instrument Guidance (CAIG); Ultrasound-CT Fusion; Image Fusion; Clear Guide SCENERGY; Needle path; Needle Guidance; CT; Ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Ultrasound-CT Fusion Guidance (Experimental): The participants in this group (test group) will utilize the ultrasound-CT fusion system for guiding needle placement.
  Interventions: Device: Ultrasound-CT Fusion
- CT Guidance (No Intervention): The participants in this group (control group) will receive the procedure with traditional CT methods and equipment, for guiding needle placement.

INTERVENTIONS:
Device: Ultrasound-CT Fusion — The Clear Guide SCENERGY is an Ultrasound-CT fusion device which supplements existing ultrasound and CT capabilities. The participants randomly selected (out of 20 patients) for use of the Clear Guide SCENERGY (test group) will receive ultrasound-CT fusion guidance from the MDs performing the procedure.
  Other Names: Clear Guide SCENERGY
  Arms: Ultrasound-CT Fusion Guidance

SUMMARY:
The objective of this research is to use the Clear Guide SCENERGY technology, an FDA approved Ultrasound-CT fusion imaging system, that allows the user to fuse CT images onto a real-time ultrasound that is being performed on the patient. This fusion system will be used to perform ultrasound guided needle placements for patients undergoing percutaneous CT guided needle-based intervention. This study will consist of 20 patients, 10 patients using the CGM SCENERGY US-CT system and 10 patients using guidance only. The primary goal of the study is to prove that the new imaging fusion system is comparable to using either CT or US guidance alone to guide needle placement.

DETAILED DESCRIPTION:
A simple 20 patient study will be performed using the CG SCENERGY system. This fusion system will be used to perform image guided needle placements for patients undergoing percutaneous CT guided needle-based intervention (CT guided biopsy, CT guided drain placement within the abdomen or pelvis, and CT guided injection of muscle or nerve within the pelvis). Only patients who are already scheduled for a CT guided procedure will be screened. The study design is as follows:

* 10 patients will have their procedure performed using the CGM SCENERGY US-CT fusion system and 10 patients will have their procedure performed using CT guidance only.
* Proper informed consent will be obtained
* Perform a CT scan with the optical adhesive skin markers in place. Markers are placed around the expected site of needle skin entry.
* The first 10 patients Group#1 (1-10) will be assigned to using the SCENERGY fusion system to complete the needle placement, and the next 10 patients Group #2 (11-20) will be assigned of continuing with CT guidance only to complete the needle placement.
* If in Group #1, the procedure will proceed as usual using the SCENERGY system to guide the needle to target. If in the Group #2, CT guidance will be used to place the needle to target.
* Once the needle is at the target, a confirmatory CT will be performed.

  * If the target is reached (i.e., the software directed the interventional radiologist to the right place, e.g. for correctly biopsying a lesion), the trial is considered a "success" and the procedure continues as normal.
  * If the needle is not in the right place, the trial is considered a "failure", and the procedure continues as normal without using the CGM software any further.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing percutaneous CT guided needle-based intervention (CT guided biopsy, CT guided drain placement within the abdomen or pelvis, and CT guided injection of muscle or nerve within the pelvis)
* Able to give written informed consent

Exclusion Criteria:

* Unable to give informed consent
* Patients undergoing CT guided needle-based interventions other than the procedures mentioned in the inclusion criteria
* Prisoners, pregnant women, and children

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-06-22 (Actual); Primary Completion 2018-06-22 (Estimated); Study Completion 2018-06-22 (Estimated)

PRIMARY OUTCOMES:
Number of CT scans or CT fluoroscopic images | Immediately following intervention (within 2 hours)

SECONDARY OUTCOMES:
Total procedure time | Immediately following intervention (within 2 hours)
  Time from the first CT scan until the needle is at the target
Time to target | Immediately following intervention (within 2 hours)
  Time from needle entering the skin until the needle is at the target
Success of needle placement | Immediately following intervention (within 2 hours)
  A confirmatory CT will be performed to check if the needle reached the target

CONTACTS AND LOCATIONS:
Overall Officials: Brian Holly, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States